CLINICAL TRIAL: NCT01488383
Title: Comparison of the Effect on Postpandrial Capillary Blood Glucose Between Oral Stevioside Versus Saccharin in Healthy Adults.
Brief Title: Effect of Stevioside in Postpandrial Glucose in Healthy Adults
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: not i
Sponsor: Basque Health Service (Other Government)
Responsible Party: Principal Investigator, Antxon Apiñaniz Fernández de LArrinoa, Primary health care physician, Basque Health Service
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ST-01
Record Dates: First submitted 2011-12-07; First posted 2011-12-08 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Hyperglycemia; Hypertension
Keywords: Hyperglycemia; Diabetes; Blood glucose; Hypertension; Anti hypertensive agents; Anti hypertensive drugs; Anti hypertensive
MeSH Terms: conditions — Hyperglycemia; Hypertension; Diabetes Mellitus | interventions — Saccharin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stevioside capsules 200mg (Experimental): Capsules of 200mg Stevioside
  Interventions: Drug: Purified extract of Rebaudina Stevia-Stevioside
- Sodium Saccharin 250 capsules (Active Comparator): Capsules of 250mg Saccharin
  Interventions: Drug: Sodium saccharin

INTERVENTIONS:
Drug: Purified extract of Rebaudina Stevia-Stevioside — volunteers will take only one capsule of stevioside (one day), and then corresponding measurements will be performed.
  Other Names: Gycostevia-95
  Arms: Stevioside capsules 200mg
Drug: Sodium saccharin — Volunteers will take one capsule of saccharin 250mg (one day) and then, corresponding measurements will be performed
  Other Names: Saccharin
  Arms: Sodium Saccharin 250 capsules

SUMMARY:
A natural sweetener (Stevia Rebaudina Bertoni) reduces blood glucose levels and blood pressure according to various preclinical and clinical studies conducted worldwide. Since it is not found many studies in the literature wich compares Stevia Rebaudiana with saccharin, we've proposed a randomized crossover clinical trial comparing the effects on postprandial capillary blood glucose and blood pressure in healthy adults.

Sample: healthy professionals from two health centers in Alava (Kakuabizkarra primary care center and Txagorritxu hospital). Inclusion criteria: Professionals of two health centers of Álava (Lakuabizkarra and Txagorritxu) and active employment status at the beginning of the trial, weighing more than 50kg and age over 18 years.

Intervention: 200mg capsules of Stevia or 250mgcapsules of saccharin. Measurements: Capillary blood glucose and blood pressure, fasting and after eating. Evaluation of satiety, hunger and fullness by questionnaire after intake, and at the end of the day.

Statistical analysis: Compare the postprandial capillary glucose levels between 8 am and 1 st hour, 2nd hour 3rd hour after intake between treatments by ANCOVA. We will also compare blood pressure before and after intake between treatments. We will also compare by t test or paired Wilcoxom (depending on the nature of the variable) the results of the questionnaire after intake between treatments.

DETAILED DESCRIPTION:
State of the art: Excessive intake of calories and sugar diets cause weight gain and impaired glucose tolerance in healthy subjects (1). These diets raise postpandrial blood glucose and insulin levels and cause metabolic and hormonal changes that induce feelings of hunger and fat deposition. These diets are also associated with diseases such as diabetes, cardiovascular disease and cancer (2).

The origin of the artificial sweeteners dates back to 1879 with the accidental discovery of saccharin. France in 1902 and the United States in 1912 officially banned its use because of their lack of nutritional value. But Europe allowed the use of saccharin during sugar rationing in the world wars (3). In the past three decades has increased the consumption of these sweeteners as it has allowed many people suffering from obesity and / or diabetes restore some degree of palatability to foods (4).

Stevia rebaudiana Bertoni (Bertoni), common name "sweet herb of Paraguay" is a plant native to Paraguay and Brazil, known by Indians as Ka'a-he'e (sweet grass). Its leaves were used since pre-Columbian times for medicinal purposes and as a sweetener because of its sweet taste (5). Japan and Brazil have more than 20 years using it as a natural sweetener. The main sweet component of Stevia is the Stevioside, a glycoside 300 times sweeter than sucrose (7).

The benefits of stevia as a dietary supplement in humans are many: it is stable, non-caloric and offers a good dental health. In addition, no significant adverse effects have occurred from their use (6).

There have been several studies that compare the decline in blood glucose and insulin levels of Stevia versus many sweeteners. It has been administered to healthy and diabetic rats (8), healthy humans (9,10), obese (10) and diabetic (11).

Another therapeutic properties of Stevia rebaudiana is a reduction in blood pressure, systolic and diastolic as Chan et al demonstrated in a randomized clinical trial conducted in China (12,13).

Toxicity studies in animals (14) and pregnant (15) have concluded that consumption of Stevia is safe at commonly used doses of sweetener (7). Furthermore, the quality of life did not deteriorate (12) nor adverse effects have been detected (16).

The available data suggest that stevia has immunostimulatory activity and inflammation modulating. But these effects have not been demonstrated in a robust in animal models or cell lines. If confirmed, the used of stevia could cause problems in some subgroups of population like in people with autoimmune diseases or gastrointestinal tract inflammation (6).

In USA it is used as a dietary supplement since 1995, but was evaluated as a sweetener by the European Scientific Committee on Food for 1984, 1989 and 1999 and concluded that it was not toxicologically acceptable because there were not enough studies (6). However, recently, the FDA, WHO and FAO have approved Stevia as a "food additive" for use in people of all ages (17).

In summary, the literature indicates that steviol can be used safely as a sweetener in the healthy population, and brings significant benefits for controlling blood glucose levels and blood pressure. However, to date there are few studies comparing Stevia with other common sweeteners. For this reason, and to compare the effect of saccharin versus Stevioside, we plan to conduct this randomized crossover clinical trial.

Study justification: Diets high in sucrose promote weight gain, causing alterations in glucose tolerance in healthy subjects (1) and are associated with metabolic disorders like diabetes wich is characterized by plasma glucose levels above the normal limits and if it isn't adequately treated can lead to complications such as neuropathy, retinopathy, neuropathy, diabetic microangiopathy and atherosclerosis.

Since diabetic patients should not eat sugar, artificial sweetener use has increased over the past three decades due to the fact that consumption of these substances has allowed many people suffering from obesity and /or diabetes to restore some degree of palatability to food (4). Among them, a natural sweetener, Stevioside also reduces the levels of postprandial glucose and insulin, and blood pressure. Besides the consumption of Stevia is safe at doses normally used as a sweetener

According to the reviewed literature, Stevioside can be used safely as a sweetener in the healthy population, providing significant benefits for controlling blood glucose levels and blood pressure with no serious adverse reactions. In the most of studies from literature, Stevioside's effect is compared with placebo, however, to date few studies have been conducted wich compare it with other sweeteners commonly used by people. For this reason, and to compare the effect and safety of Stevioside versus Saccharin we have planed this randomized crossover clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Professionals of sanitary centers in active working situation at start date of clinical trial.
* Weight over 50kg.
* Age over 18 years.

Exclusion Criteria:

* History of diabetes mellitus, arterial hypertension or hypercholesterolemia.
* Obesity (BMI ≥ 30kg/m2)
* Cardiovascular disease.
* Enrollment in other clinical trial with medicaments within three months.
* Any endocrine disease other than diabetes.
* Glucocorticoids treatment.
* Pregnant women.
* Herball allergy.
* Autoimmune diseases.
* Inflammatory bowel disease.
* Allergy to sulfonamides.
* Steven-Johnson syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-09; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
change in capillary blood glucose levels | at baseline and and at first hour after intake
  Change in capillary blood glucose levels after treatment

SECONDARY OUTCOMES:
change in blood pressure | at baseline and and at third hour after intake
  Change in blodd pressure after treatment
feeling of fullness, hunger and satiety after intake | At baseline and and at third hour after intake
  feeling of fullness, hunger and satiety after treatment
Adverse reactions of treatments (nausea, diarrhea, vomiting, allergic signs) | After intake
  To describe and compare the adverse reactions of each treatment nausea, diarrhea, vomiting, allergic signs.

CONTACTS AND LOCATIONS:
Locations (1):
- Basque Public Health Service-Osakidetza (Lakuabizkarra primary care center and Txagorritxu hospital), Vitoria-Gasteiz, Alava, Spain